CLINICAL TRIAL: NCT02225587
Title: Sequential Administration of Prevnar 13™ and Pneumovax™ 23 in Healthy Subjects 50 Years of Age and Older
Brief Title: Evaluation of the Safety and Immunogenicity of Sequential Administration of Prevnar 13™ and Pneumovax™ 23 in Healthy Participants 50 Years of Age and Older (V110-029)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V110-029; 2013-003027-11 (EudraCT Number); V110-029 (Other: Merck)
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo (Experimental): Prevnar 13™ 0.5 mL intramuscular injection on Day 1, Pneumovax™ 23 0.5 mL intramuscular injection at Week 8, and Placebo 0.5 mL intramuscular injection at Week 26. Injections are to be administered in alternating limbs, if possible.
  Interventions: Biological: Prevnar 13™; Biological: Pneumovax™ 23; Biological: Placebo
- Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23 (Placebo Comparator): Prevnar 13™ 0.5 mL intramuscular injection on Day 1, Placebo 0.5 mL intramuscular injection at Week 8, and Pneumovax™ 23 0.5 mL intramuscular injection at Week 26. Injections are to be administered in alternating limbs, if possible.
  Interventions: Biological: Prevnar 13™; Biological: Pneumovax™ 23; Biological: Placebo

INTERVENTIONS:
Biological: Prevnar 13™ — Pneumococcal vaccine containing serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F. Injections are to be administered into the deltoid muscle of the upper arm.
Biological: Pneumovax™ 23 — Pneumococcal vaccine containing serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F. Injections are to be administered into the deltoid muscle of the upper arm.
Biological: Placebo — Injections are to be administered into the deltoid muscle of the upper arm.

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of sequential administration of Prevnar 13™ and Pneumovax™ 23 in healthy participants 50 years of age and older. The primary hypotheses in the study are that 1) geometric mean titers (GMTs) to pneumococcal serotypes 22F and 33F (serotypes in Pneumovax™ 23 but not in Prevnar 13™) as measured at Week 12 are superior in participants administered Prevnar 13™ on Day 1 and Pneumovax™ 23 at Week 8, as compared with participants administered Prevnar 13™ on Day 1 and placebo at Week 8 and 2) GMTs to pneumococcal serotypes shared by the two vaccines as measured at Week 12 are non-inferior in participants administered Prevnar 13™ followed by Pneumovax™ 23 as compared with participants administered Prevnar 13™ followed by placebo.

ELIGIBILITY:
Inclusion Criteria:

* Any chronic illness must be documented to be in stable condition
* Male, or a female agrees to remain abstinent, or use, or have their partner use, 2 acceptable methods of contraception through 6 weeks after receiving study vaccination; or a female who is not of reproductive potential

Exclusion Criteria:

* Is or has an immediate family member who is investigational site or sponsor staff directly involved with this trial
* Prior administration of any pneumococcal vaccine
* History of invasive pneumococcal disease
* Known hypersensitivity to any component of the pneumococcal polysaccharide vaccine, of the pneumococcal conjugate vaccine, or any diphtheria toxoid-containing vaccine
* Known or suspected impairment of immunological function, documented Human Immunodeficiency Virus (HIV) infection, asplenia, or history of autoimmune disease
* Received systemic corticosteroids (equivalent of >=2 mg/kg total daily dose of prednisone or >=20 mg/kg for persons weighing >10 kg) for >=14 consecutive days and has not completed treatment <=30 days before study vaccination, or has received systemic corticosteroids exceeding physiological doses (~5 mg/day prednisone equivalent) within 14 days before study vaccination (topical, ophthalmic, intra-articular, and inhaled/nebulized steroids are permitted).
* Has a coagulation disorder contraindicating intramuscular vaccination
* Receiving immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and treatments associated with organ or bone marrow transplantation or autoimmune disease
* Received a blood transfusion or blood products, including immunoglobulins <=6 months before receiving study vaccine, or is scheduled to receive them within 30 days
* Participated in another clinical study of an investigational product <=2 months before or during the current study
* Is breast-feeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2015-07-06 (Actual); Study Completion 2015-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Buchwald UK, Andrews CP, Ervin J, Peterson JT, Tamms GM, Krupa D, Ajiboye P, Roalfe L, Krick AL, Sterling TM, Wang M, Martin JC, Stek JE, Kohn MA, Folaranmi T, Abeygunawardana C, Hartzel J, Musey LK; V110-029 Study Group. Sequential administration of Prevnar 13 and PNEUMOVAX 23 in healthy participants 50 years of age and older. Hum Vaccin Immunother. 2021 Aug 3;17(8):2678-2690. doi: 10.1080/21645515.2021.1888621. Epub 2021 May 21. PMID 34019468

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo: Prevnar 13™ 0.5 mL intramuscular injection on Day 1, Pneumovax™ 23 0.5 mL intramuscular injection at Week 8, and Placebo 0.5 mL intramuscular injection at Week 26. Injections were administered in alternating limbs.
- Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23: Prevnar 13™ 0.5 mL intramuscular injection on Day 1, Placebo 0.5 mL intramuscular injection at Week 8, and Pneumovax™ 23 0.5 mL intramuscular injection at Week 26. Injections were administered in alternating limbs.
Period: Overall Study
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Started (Received Vaccination 1) | 200 | 200
Vaccination 2 (Received Vaccination 2) | 188 | 185
Vaccination 3 (Received Vaccination 3) | 172 | 164
Completed | 172 | 162
Not Completed | 28 | 38
Not completed — Adverse Event | 5 | 5
Not completed — Lost to Follow-up | 5 | 5
Not completed — Non-Compliance With Study Drug | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Participant Moved | 1 | 0
Not completed — Withdrawal by Subject | 13 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23 | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.6) | 64.2 (8.9) | 64.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 107 | 219
  Male | 88 | 93 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 35 | 75
  Not Hispanic or Latino | 158 | 164 | 322
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 23 | 37
  White | 176 | 163 | 339
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 14 days after any vaccination (Up to 28 weeks)
Population: Participants who received at least 1 dose of treatment and followed up for safety. Two participants from Group 1, and 1 participant from Group 2 were not analyzed due to lack of follow-up data. As the objective was to report the combined safety of the two vaccines given 8 or 26 weeks apart, results are presented for the sequence of vaccinations.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 198 | 199
Percentage of participants | 89.9 | 84.4

2. Primary Outcome: Percentage of Participants With an Injection-site Adverse Event
Description: An injection site adverse event (AE) includes the following AEs at the injection site: redness, swelling, and pain/tenderness.
Time Frame: Up to 14 days after any vaccination (Up to 28 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 198 | 199
Percentage of participants | 86.4 | 77.9

3. Primary Outcome: Percentage of Participants With a Systemic Adverse Event
Description: Systemic adverse events (AEs) include, but are not restricted to the following AE terms: muscle pain, joint pain, headache, and tiredness.
Time Frame: Up to 14 days after any vaccination (Up to 28 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 198 | 199
Percentage of participants | 76.8 | 74.4

4. Primary Outcome: Percentage of Participants With a Serious Adverse Event (SAE)
Description: A serious adverse event (SAE) is any adverse event occurring at any dose or during any use of Sponsor's product that: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is another important medical event; is a cancer; or is associated with an overdose.
Time Frame: Up to 30 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 198 | 199
Percentage of participants | 4.5 | 5.5

5. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event (SAE) or Vaccine-related Death
Description: A serious adverse event (SAE) is any adverse event occurring at any dose or during any use of Sponsor's product that: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is another important medical event; is a cancer; or is associated with an overdose. The investigator determined whether the SAE or death was related to vaccine treatment.
Time Frame: Up to 30 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 198 | 199
Percentage of participants | 0 | 0

6. Primary Outcome: Percentage of Participants Who Discontinued Vaccination Due to an Adverse Event
Description: as for outcome 1
Time Frame: Up to 26 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 198 | 199
Percentage of participants | 2.5 | 2.5

7. Primary Outcome: Geometric Mean Titers to Pneumococcal Serotypes 22F and 33F at Week 12
Description: Vaccine-induced functional antibodies to serotypes 22F and 33F, which are unique to PNEUMOVAX™ 23, were measured by the multiplex opsonophagocytic activity 4 (MOPA-4) assay, which is based on the ability of antibody in the serum to initiate killing of bacterial pneumococci.
Time Frame: Week 12
Population: All randomized participants who received at least 1 vaccination and provided serology data for the particular serotype tested; with appropriate day ranges for vaccinations and blood draws, and excludes participants with important deviations from the protocol that may substantially affect the results.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 172 | 172
Titer
  Serotype 22F: number analyzed (Participants) | 166 | 157
  Serotype 22F | 1766.3 [1303.2 to 2394.1] | 39.0 [28.3 to 53.7]
  Serotype 33F | 10413.0 [8178.9 to 13257.4] | 1189.9 [898.6 to 1575.6]

8. Primary Outcome: Geometric Mean Titers to Pneumococcal Serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F, at Week 12
Description: Vaccine-induced functional antibodies to serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F, which are contained in both Prevnar 13™ and PNEUMOVAX™ 23, were measured by the MOPA-4 assay, which is based on the ability of antibody in the serum to initiate killing of bacterial pneumococci.
Time Frame: Week 12
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 172 | 179
Titer
  Serotype 1: number analyzed (Participants) | 168 | 173
  Serotype 1 | 81.7 [60.4 to 110.7] | 57.1 [41.1 to 79.3]
  Serotype 3: number analyzed (Participants) | 151 | 155
  Serotype 3 | 43.4 [33.7 to 55.9] | 17.5 [13.5 to 22.5]
  Serotype 4: number analyzed (Participants) | 171 | 176
  Serotype 4 | 1079.3 [885.7 to 1315.2] | 780.0 [629.1 to 967.1]
  Serotype 5: number analyzed (Participants) | 171 | 178
  Serotype 5 | 198.6 [145.6 to 271.0] | 148.4 [107.9 to 204.1]
  Serotype 6B: number analyzed (Participants) | 170 | 179
  Serotype 6B | 1956.9 [1575.3 to 2431.0] | 1148.1 [889.0 to 1482.6]
  Serotype 7F | 2250.8 [1889.3 to 2681.5] | 1751.8 [1422.4 to 2157.6]
  Serotype 9V: number analyzed (Participants) | 164 | 175
  Serotype 9V | 1472.3 [1190.9 to 1820.2] | 1017.6 [790.8 to 1309.4]
  Serotype 14: number analyzed (Participants) | 172 | 178
  Serotype 14 | 2106.8 [1689.6 to 2627.0] | 1945.0 [1572.9 to 2405.1]
  Serotype 18C: number analyzed (Participants) | 171 | 175
  Serotype 18C | 2101.9 [1732.6 to 2550.0] | 1587.1 [1259.1 to 2000.5]
  Serotype 19A | 1785.8 [1506.1 to 2117.6] | 1425.9 [1164.7 to 1745.8]
  Serotype 19F: number analyzed (Participants) | 171 | 178
  Serotype 19F | 1051.0 [862.1 to 1281.3] | 627.2 [490.5 to 802.2]
  Serotype 23F: number analyzed (Participants) | 164 | 176
  Serotype 23F | 1155.6 [867.2 to 1539.9] | 716.9 [521.1 to 986.3]

9. Secondary Outcome: Geometric Mean Titers to Pneumococcal Serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F at Week 8
Description: Vaccine-induced functional antibodies were measured by the MOPA-4 assay, which is based on the ability of antibody in the serum to initiate killing of bacterial pneumococci.
Time Frame: Week 8
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 43 | 47
Titer
  Serotype 1: number analyzed (Participants) | 42 | 44
  Serotype 1 | 100.7 [50.5 to 200.9] | 54.7 [27.5 to 108.5]
  Serotype 3: number analyzed (Participants) | 39 | 45
  Serotype 3 | 52.8 [32.2 to 86.5] | 27.8 [16.6 to 46.5]
  Serotype 4: number analyzed (Participants) | 43 | 46
  Serotype 4 | 1075.7 [671.4 to 1723.5] | 1051.0 [696.0 to 1587.0]
  Serotype 5 | 350.5 [193.2 to 636.1] | 143.9 [77.7 to 266.3]
  Serotype 6A | 3945.3 [2301.9 to 6762.2] | 4024.1 [2622.8 to 6174.1]
  Serotype 6B: number analyzed (Participants) | 42 | 47
  Serotype 6B | 2154.2 [1325.4 to 3501.3] | 1259.7 [707.3 to 2243.5]
  Serotype 7F | 3830.5 [2654.6 to 5527.2] | 2064.0 [1287.4 to 3309.0]
  Serotype 9V | 1555.6 [988.7 to 2447.6] | 1606.5 [1064.5 to 2424.6]
  Serotype 14: number analyzed (Participants) | 42 | 46
  Serotype 14 | 2417.0 [1547.8 to 3774.1] | 1586.4 [901.6 to 2791.3]
  Serotype 18C | 1890.8 [1313.3 to 2722.1] | 1563.7 [857.8 to 2850.3]
  Serotype 19A: number analyzed (Participants) | 43 | 46
  Serotype 19A | 2102.3 [1567.6 to 2819.5] | 1819.8 [1300.2 to 2547.0]
  Serotype 19F: number analyzed (Participants) | 43 | 46
  Serotype 19F | 1039.4 [646.0 to 1672.2] | 640.4 [378.1 to 1084.9]
  Serotype 22F: number analyzed (Participants) | 42 | 43
  Serotype 22F | 116.4 [54.9 to 246.8] | 30.9 [16.6 to 57.5]
  Serotype 23F: number analyzed (Participants) | 43 | 46
  Serotype 23F | 1245.8 [656.9 to 2362.5] | 779.8 [414.3 to 1467.8]
  Serotype 33F: number analyzed (Participants) | 42 | 47
  Serotype 33F | 1515.4 [914.3 to 2511.5] | 1984.0 [1207.9 to 3259.0]

10. Secondary Outcome: Geometric Mean Titers to Pneumococcal Serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F at Week 26
Description: as for outcome 9
Time Frame: Week 26
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 44 | 48
Titer
  Serotype 1: number analyzed (Participants) | 43 | 48
  Serotype 1 | 39.7 [20.4 to 77.4] | 18.9 [10.7 to 33.3]
  Serotype 3: number analyzed (Participants) | 34 | 43
  Serotype 3 | 19.6 [12.0 to 32.1] | 9.2 [6.2 to 13.7]
  Serotype 4: number analyzed (Participants) | 42 | 47
  Serotype 4 | 737.1 [451.9 to 1202.1] | 788.4 [535.3 to 1161.1]
  Serotype 5: number analyzed (Participants) | 43 | 46
  Serotype 5 | 114.4 [58.5 to 223.4] | 65.6 [36.2 to 118.8]
  Serotype 6A: number analyzed (Participants) | 42 | 47
  Serotype 6A | 1843.2 [1111.0 to 3057.8] | 1152.9 [655.0 to 2029.3]
  Serotype 6B: number analyzed (Participants) | 44 | 45
  Serotype 6B | 1157.0 [639.0 to 2094.7] | 1125.1 [689.7 to 1835.6]
  Serotype 7F | 1204.9 [832.1 to 1744.8] | 770.7 [499.5 to 1189.2]
  Serotype 9V: number analyzed (Participants) | 42 | 45
  Serotype 9V | 698.2 [437.7 to 1113.8] | 806.5 [500.9 to 1298.7]
  Serotype 14: number analyzed (Participants) | 43 | 47
  Serotype 14 | 1458.2 [949.2 to 2240.1] | 1373.9 [879.5 to 2146.1]
  Serotype 18C: number analyzed (Participants) | 44 | 45
  Serotype 18C | 914.2 [594.3 to 1406.2] | 691.1 [383.1 to 1246.7]
  Serotype 19A: number analyzed (Participants) | 43 | 48
  Serotype 19A | 1024.3 [749.4 to 1400.1] | 806.3 [539.3 to 1205.6]
  Serotype 19F: number analyzed (Participants) | 43 | 47
  Serotype 19F | 563.7 [344.0 to 923.7] | 228.9 [126.1 to 415.5]
  Serotype 22F: number analyzed (Participants) | 41 | 45
  Serotype 22F | 1228.3 [733.3 to 2057.4] | 45.2 [23.5 to 86.7]
  Serotype 23F: number analyzed (Participants) | 43 | 46
  Serotype 23F | 653.8 [315.8 to 1353.4] | 366.6 [195.9 to 685.9]
  Serotype 33F: number analyzed (Participants) | 44 | 46
  Serotype 33F | 4672.8 [2968.8 to 7354.7] | 1151.4 [660.4 to 2007.6]

11. Secondary Outcome: Geometric Mean Titers to Pneumococcal Serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F at Week 30
Description: as for outcome 9
Time Frame: Week 30
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
Number analyzed (Participants) | 88 | 94
Titer
  Serotype 1: number analyzed (Participants) | 86 | 89
  Serotype 1 | 36.0 [23.2 to 55.9] | 43.4 [28.8 to 65.5]
  Serotype 3: number analyzed (Participants) | 77 | 86
  Serotype 3 | 13.9 [10.2 to 18.9] | 32.8 [23.8 to 45.2]
  Serotype 4: number analyzed (Participants) | 87 | 93
  Serotype 4 | 803.6 [601.2 to 1074.2] | 1060.0 [796.2 to 1411.3]
  Serotype 5: number analyzed (Participants) | 87 | 93
  Serotype 5 | 81.5 [51.1 to 130.0] | 117.3 [83.5 to 164.9]
  Serotype 6A: number analyzed (Participants) | 85 | 91
  Serotype 6A | 1673.9 [1141.5 to 2454.5] | 1782.7 [1255.1 to 2532.1]
  Serotype 6B: number analyzed (Participants) | 84 | 92
  Serotype 6B | 1330.3 [911.8 to 1940.8] | 1343.6 [993.3 to 1817.3]
  Serotype 7F: number analyzed (Participants) | 87 | 93
  Serotype 7F | 877.7 [683.3 to 1127.5] | 1248.4 [955.3 to 1631.4]
  Serotype 9V: number analyzed (Participants) | 87 | 93
  Serotype 9V | 628.9 [444.3 to 890.4] | 1134.8 [841.4 to 1530.5]
  Serotype 14: number analyzed (Participants) | 87 | 93
  Serotype 14 | 1762.9 [1257.3 to 2471.7] | 1963.3 [1441.9 to 2673.4]
  Serotype 18C: number analyzed (Participants) | 88 | 92
  Serotype 18C | 779.3 [582.9 to 1041.8] | 1125.6 [843.5 to 1502.1]
  Serotype 19A: number analyzed (Participants) | 87 | 94
  Serotype 19A | 845.5 [649.5 to 1100.6] | 1256.1 [1027.9 to 1535.0]
  Serotype 19F: number analyzed (Participants) | 88 | 93
  Serotype 19F | 349.1 [236.9 to 514.5] | 880.8 [663.9 to 1168.6]
  Serotype 22F: number analyzed (Participants) | 81 | 92
  Serotype 22F | 1124.7 [751.7 to 1682.9] | 982.1 [642.6 to 1501.0]
  Serotype 23F: number analyzed (Participants) | 86 | 93
  Serotype 23F | 574.3 [367.6 to 897.2] | 755.6 [521.6 to 1094.4]
  Serotype 33F: number analyzed (Participants) | 86 | 94
  Serotype 33F | 5917.9 [4199.6 to 8339.4] | 7853.5 [5521.3 to 11171.0]

ADVERSE EVENTS:
Time Frame: Up to 30 Weeks
Description: Participants who received at least 1 dose of study intervention. Adverse Events, including injection specific Adverse Events, were pre-specified to be monitored/assessed per vaccination sequence group, and are therefore reported per vaccination sequence group..
Arm/Group | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23
All-Cause Mortality (participants affected / at risk) | 1/200 | 0/200
Serious Adverse Events (participants affected / at risk) | 9/200 | 11/200
Other Adverse Events (participants affected / at risk) | 177/200 | 165/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo (N=200) | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23 (N=200)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Prevnar 13™ → Pneumovax™ 23 → Placebo (N=200) | Group 2: Prevnar 13™ → Placebo → Pneumovax™ 23 (N=200)
Fatigue (General disorders) | 100 (209) | 89 (159)
Injection site erythema (General disorders) | 99 (138) | 72 (93)
Injection site pain (General disorders) | 168 (357) | 151 (289)
Injection site swelling (General disorders) | 111 (173) | 78 (111)
Arthralgia (Musculoskeletal and connective tissue disorders) | 58 (105) | 55 (80)
Myalgia (Musculoskeletal and connective tissue disorders) | 123 (210) | 115 (184)
Headache (Nervous system disorders) | 78 (140) | 60 (114)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.